CLINICAL TRIAL: NCT04923048
Title: A Phase Ⅰ/Ⅱ, Open-Label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of GB261 in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: A Safety, Tolerability, Pharmacokinetics and Efficacy Study of GB261 in B-Cell NHL and CLL.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB261-001
Record Dates: First submitted 2021-06-04; First posted 2021-06-11 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2022-06

CONDITIONS: B Cell NHL; CLL
Keywords: B cell NHL, Phase 1/2,GB261,bispecific antibody,CD20/CD3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB261 (Experimental): Participants will receive GB261 via intravenous (IV) infusion as a single agent on Day 1, Day 8 and Day 15 of Cycle 1 and 2 followed by Day 1 of each cycle（21 days per cycle） afterwards until disease progression or other situations specified in the protocol, whichever comes earlier.
  Interventions: Biological: GB261

INTERVENTIONS:
Biological: GB261 — Drug:GB261 IV, participants with B-cell NHL or CLL will receive GB261 via IV infusion weekly for the first two cycles(1cycle=21days), followed by Q3W from C3 and afterwards in given doses until progression disease or other situations specified in the protocol, whichever comes earlier.

SUMMARY:
This is a Phase 1/2 study of GB261 in participants with relapsed or refractory B-cell NHL and CLL. The study will consist of a dose-escalation stage(Phase 1), an expansion stage(Phase 2a) and Phase 2b stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
2. CD20+ B-cell Non-Hodgkin Lymphoma or CLL who have relapsed or failed to respond to at least one prior treatment regimen and for whom there is no available therapy expected to improve survival
3. Adequate hepatic, hematologic, and renal function

Exclusion Criteria:

1. Burkitt lymphoma, lymphoplasmacytic lymphoma or B lymphoblastic leukemia
2. Prior treatment with systemic anti-lymphoma therapy within 4 weeks or five half-lives of the drug (which is shorter) prior to the first GB261 infusion
3. History of auto-SCT or CAR-T therapy in the past 180 days and/or with any of protocol specified conditions
4. Prior allo-SCT or allogeneic CAR-T
5. Prior solid organ transplantation
6. Autoimmune disease with the exceptions specified in the protocol
7. History of central nervous system(CNS) lymphoma or other CNS disease
8. Significant cardiovascular or pulmonary disease
9. Hepatitis B or C or human immunodeficiency virus (HIV)
10. Pregnant or lactating or intending to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | During Cycle 1 (up to 21 days)
Dose Limiting Toxicity | During Cycle 1 (up to 21 days)
Percentage of participants with adverse events | From first dosing until 90 days after the last treatment
Objective Response Rate | Through study completion, an average of 3 years

SECONDARY OUTCOMES:
Cmax | At predefined intervals up to 106 days
Tmax | At predefined intervals up to 106 days
Area Under the Curve | At predefined intervals up to 106 days
t1/2 | At predefined intervals up to 106 days
Clearance | At predefined intervals up to 106 days
Vz | At predefined intervals up to 106 days
Anti-Drug Antibody | At predefined intervals up to 3 years
Progression Free Survival | Through study completion, an average of 3 years
Duration of Objective Response | Through study completion, an average of 3 years
Duration of Objective Complete Response | Through study completion, an average of 3 years
Overall Survival | Through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - St Vincent's Hospital/The Kinghorn Cancer Centre, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Cabrini hospital, Melbourne, The State of Victoria
  - Alfred hospital, Melbourne, The State of Vitoria
  - Peninsula & South Eastern Haematology & Oncology Group, Melbourne, The State of Vitoria
  - One Clinical Research Pty Ltd, Mount Pleasant, Western Australia

IPD SHARING:
Plan to Share IPD: No